CLINICAL TRIAL: NCT04077216
Title: Effect of Extra Virgin Olive Oil on Postprandial Blood Glucose in Type 2 Diabetes Mellitus: A Randomized Controlled Trial
Brief Title: Effect of Extra Virgin Olive Oil on Postprandial Blood Glucose in Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makati Medical Center (Other)
Responsible Party: Principal Investigator, Daphne Gayle P Galang, Fellow, Section of Endocrinology, Department of Internal Medicine, Makati Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: MakatiMedCtr
Record Dates: First submitted 2019-08-29; First posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus Type 2; Diet therapy; Extra virgin olive oil
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Crossover trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Initially received the test meal with EVOO, then on crossover, received the meal without EVOO
  Interventions: Dietary Supplement: Extra Virgin Olive Oil (EVOO)
- Group B (No Intervention): Initially received the test meal without EVOO, then on crossover, received the meal without EVOO

INTERVENTIONS:
Dietary Supplement: Extra Virgin Olive Oil (EVOO) — This study used the FDA approved Doña Elena Extra virgin olive oil, which is readily available in local supermarkets. Its free acidity expressed as oleic acid was found to be 0.26%, comparable with the International food standards.15
  Arms: Group A

SUMMARY:
Extra virgin olive oil (EVOO) is known for its cardiovascular effects and its effect on glucose lowering. However, the effects of EVOO on the blood glucose of Type 2 Diabetes Mellitus Filipino patients has not been studied. The investigators aimed to determine whether a significant difference exists in meals containing EVOO versus meals without EVOO among Type 2 Diabetes Mellitus patients.

Thirteen patients were included in this randomized controlled cross-over trial. They were randomized to receive a meal with or without EVOO followed by a one week wash out period, where they were given the other intervention. The primary outcome is the trans-meal blood glucose, which is calculated as the percent change in 2-hour postprandial blood glucose.

DETAILED DESCRIPTION:
During their first visit, the participants were oriented on the conduct of the study. They were advised to be compliant with their medications throughout the duration of the trial.

On their second visit, participants were asked to do a six to eight-hour overnight fast, and their fasting blood sugar was drawn. Serum samples were analyzed through the hexokinase method. The participants were then randomly allocated (first allocation) by the dietician through a coin toss to receive a standard breakfast without EVOO or a meal admixed with one tablespoon of EVOO. The standard meals were labeled with serial numbers, and both the participants and the investigator were blinded to the intervention. The meals were consumed steadily in 15 to 20 minutes, after which, the food containers were collected to ensure its full consumption. Breakfast was chosen in order to avoid a second meal bias. The participants were asked to sit in the waiting area of the laboratory until the 2-hour postprandial blood sugar was due to be drawn.

After a one-week washout period, the participants were asked to come back for a cross over to the other treatment arm (second allocation). The participants were given the same test meal to ensure that that the glycemic index of the food remained constant.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged 30-65 years old
2. diagnosed with Type 2 Diabetes Mellitus
3. body mass index under the overweight or obese class I category (by Asia Pacific guidelines)

Exclusion Criteria:

1. pregnant patients
2. patients with history of frequent hypoglycemic episodes
3. those at high risk of developing ketoacidosis and hyperglycemic hyperosmolar syndrome
4. those with identified acute stress during the study (illness, fever, trauma leading to hospitalization)
5. current intake of steroids
6. olive oil allergy or intolerance
7. digestive disorders

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
trans-meal blood glucose | 2 hours
  percent change in 2-hour postprandial blood glucose. This was calculated as the fasting blood sugar subtracted from the 2-hour postprandial glucose divided by the fasting blood sugar multiplied by 100

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jocelyn Capuli-Isidro, MD, Principal Investigator — Makati Medical Center; Ma. Cecilia Gonzales, MD, Principal Investigator — Makati Medical Center; Andrea Marie Macabuag-Oliva, MD, Principal Investigator — Makati Medical Center
Locations (1):
- Makati Medical Center, Makati City, NCR, Philippines

IPD SHARING:
Plan to Share IPD: No
Data gathered from this study were treated in conformance with the principles of confidentiality, codes were used in data collection forms and documents accessible only by the primary investigator. Explicit consent for sharing individual participant data was not taken.

REFERENCES:
- [Background] Buckland G, Gonzalez CA. The role of olive oil in disease prevention: a focus on the recent epidemiological evidence from cohort studies and dietary intervention trials. Br J Nutr. 2015 Apr;113 Suppl 2:S94-101. doi: 10.1017/S0007114514003936. PMID 26148926
- [Background] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary prevention of cardiovascular disease with a Mediterranean diet. N Engl J Med. 2013 Apr 4;368(14):1279-90. doi: 10.1056/NEJMoa1200303. Epub 2013 Feb 25. PMID 23432189 (Retraction: PMID 29897867 N Engl J Med. 2018 Jun 21;378(25):2441-2442)
- [Background] Schwingshackl L, Christoph M, Hoffmann G. Effects of Olive Oil on Markers of Inflammation and Endothelial Function-A Systematic Review and Meta-Analysis. Nutrients. 2015 Sep 11;7(9):7651-75. doi: 10.3390/nu7095356. PMID 26378571
- [Background] Violi F, Loffredo L, Pignatelli P, Angelico F, Bartimoccia S, Nocella C, Cangemi R, Petruccioli A, Monticolo R, Pastori D, Carnevale R. Extra virgin olive oil use is associated with improved post-prandial blood glucose and LDL cholesterol in healthy subjects. Nutr Diabetes. 2015 Jul 20;5(7):e172. doi: 10.1038/nutd.2015.23. PMID 26192450
- [Background] Bozzetto L, Alderisio A, Giorgini M, Barone F, Giacco A, Riccardi G, Rivellese AA, Annuzzi G. Extra-Virgin Olive Oil Reduces Glycemic Response to a High-Glycemic Index Meal in Patients With Type 1 Diabetes: A Randomized Controlled Trial. Diabetes Care. 2016 Apr;39(4):518-24. doi: 10.2337/dc15-2189. Epub 2016 Feb 9. PMID 26861923
- [Background] Holst JJ, Vilsboll T, Deacon CF. The incretin system and its role in type 2 diabetes mellitus. Mol Cell Endocrinol. 2009 Jan 15;297(1-2):127-36. doi: 10.1016/j.mce.2008.08.012. Epub 2008 Aug 20. PMID 18786605
- [Background] Evert AB, Boucher JL, Cypress M, Dunbar SA, Franz MJ, Mayer-Davis EJ, Neumiller JJ, Nwankwo R, Verdi CL, Urbanski P, Yancy WS Jr; American Diabetes Association. Nutrition therapy recommendations for the management of adults with diabetes. Diabetes Care. 2013 Nov;36(11):3821-42. doi: 10.2337/dc13-2042. Epub 2013 Oct 9. PMID 24107659
- See also: 2018 Expanded National Nutrition Survey by the Food and Nutrition Research Institute — https://www.fnri.dost.gov.ph
- See also: Trade standard applying to olive oil and olive pomace oil by the International Olive Oil Council (IOC) — http://www.internationaloliveoil.org/estaticos/view/222-standards

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT04077216/Prot_SAP_000.pdf